CLINICAL TRIAL: NCT03494257
Title: Effect of Fixed Brinzolamide-brimonidine Combination on Intraocular Pressure After Phacoemulsification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Constantinos D. Georgakopoulos, MD, PhD, Associate Professor in Ophthalmology, University Hospital of Patras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 58/15.02.2018/5104
Record Dates: First submitted 2018-04-02; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Cataract; Intraocular Pressure
Keywords: phacoemulsification; intraocular pressure; cataract; brinzolamide; brimonidinde; fixed combination
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Prospective randomized double-masked comparative study
Who Masked: Participant, Investigator
Masking Description: Patients will be unaware of their groupe assignment. The investigator who will measure the IOP will also be masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brinzolamide-Brimonidine fixed combination (Active Comparator): 1 drop of the brinzolamide-brimonidine fixed combination instilled in the patients cul de sac immediately after surgery
  Interventions: Drug: Brinzolamide-Brimonidine fixed combination
- No topical IOP reducing medication (No Intervention): No IOP reducing drops instilled after surgery

INTERVENTIONS:
Drug: Brinzolamide-Brimonidine fixed combination — Simbrinza 0.2%-1% Ophthalmic Suspension
  Other Names: Simbrinza, 0.2%-1% Ophthalmic Suspension
  Arms: Brinzolamide-Brimonidine fixed combination

SUMMARY:
This study aims to evaluate the effect of fixed brinzolamide-brimonidine combination on intaocular pressure after uncomplicated phacoemulsification surgery.

Patients scheduled for phacoemulsification will be randomly assigned to 1 of 2 groups.

The treatment group will receive 1 drop of brimonidine-brinzolamide fixed combination immediately after surgery, and the control group will receive no treatment. The IOP will be measured preoperatively and at 6, 12, and 24 hours postoperatively.

DETAILED DESCRIPTION:
Phacoemulsification with the use of an ophthalmic viscosurgical device (OVD) and implantation of a foldable intraocular lens (IOL) is the preferred technique for cataract surgery today.

OVDs in spite of their advantages in phacoemulsification surgery, have been correlated with intraocular pressure (IOP) increase within the first 24 hours postoperatively. This constitutes a frequent short-term complication of cataract surgery and can lead to corneal edema and pain. This IOP rise may also increase the risk of retinal artery occlusion, ischemic optic neuropathy, and deterioration of preexisting glaucomatous nerve damage.

DuoVisc, an OVD that consists of Viscoat (chondroitin sulfate 4.0%-sodium hyaluronate 3.0%) in combination with Provisc (sodium hyaluronate 1.0%) is the most frequently used OVD during cataract surgery.

To prevent IOP spikes postoperatively, various antiglaucoma agents have been used. Brinzolamide is a carbonic anhydrase inhibitor that acts upon the ciliary processes and reduces aqueous humor secretion.Brimonidine is a highly selective a2-adrenergic agonist that increases uveoscleral outflow and reduces aqueous humor production.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo cataract surgery by phacoemulsification.

Exclusion Criteria:

* previous ocular surgery
* ocular hypertension
* pseudoexfoliation syndrome
* pigment dispersion syndrome
* glaucoma
* history of severe cardiovascular disease, cerebral or coronary insufficiency, depression, Raynaud's phenomenon, orthostatic hypotension or thromboangiitis obliterans
* hypersensitivity to sulfonamides or brimonidine

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
IOP at 6 hours after surgery | 6 hours postoperatively
  IOP will be measured by the same Goldman applanation tonometer used preoperatively

SECONDARY OUTCOMES:
IOP at 12 hours after surgery | 12 hours postoperatively
  IOP will be measured by the same Goldman applanation tonometer used preoperatively
IOP at 24 hours after surgery | 12 hours postoperatively
  IOP will be measured by the same Goldman applanation tonometer used preoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Constantine Georgakopoulos, MD, PhD, Principal Investigator — Medical School, University of Patras, Greece
Locations (1):
- University Hospital of Patras, Pátrai, Achaia, Greece